CLINICAL TRIAL: NCT05703074
Title: The Efficacy and Safety of a Mental Intervention Program vs. Usual Care and Nicotinamide Riboside (NR) vs. Placebo for Improving Health-related Quality of Life in Long Covid: A 2 x 2 Factorial Randomized Controlled Trial
Brief Title: Mental Intervention and Nicotinamide Riboside Supplementation in Long Covid
Acronym: MINIRICO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Vegard Wyller, Professor, University Hospital, Akershus
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 983971636
Record Dates: First submitted 2023-01-25; First posted 2023-01-27 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: A 2 x 2 factorial randomized controlled trial, where Mind-Body Reprocessing Therapy (MBRT) is compared with care as usual and Nicotinamide Riboside (NR) is compared with placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For the NR vs placebo comparison, participants, care providers, investigators and outcome assessors are blinded. For the MBRT vs. usual care comparison, due to the nature of the intervention, only outcome assessors are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MBRT and NR (Other): Psychological therapy and dietary supplement
  Interventions: Dietary Supplement: Nicotinamide Riboside (NR); Behavioral: Mind-body reprocessing therapy (MBRT)
- MBRT and placebo (Other): Psychological therapy and placebo dietary supplement
  Interventions: Behavioral: Mind-body reprocessing therapy (MBRT); Dietary Supplement: Placebo
- Care as usual and NR (Other): No psychological therapy (information only) and dietary supplement
  Interventions: Dietary Supplement: Nicotinamide Riboside (NR); Behavioral: Care as usual
- Care as usual and placebo (Other): No psychological therapy (information only) and placebo dietary supplement
  Interventions: Behavioral: Care as usual; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside (NR) — 4 capsules (a total of 1000 mg) 2 times daily for 84 days
  Arms: Care as usual and NR; MBRT and NR
Behavioral: Mind-body reprocessing therapy (MBRT) — 4-6 face-to-face meetings over 3-4 weeks, unlimited access to designated online resources.
  Arms: MBRT and NR; MBRT and placebo
Behavioral: Care as usual — A brief self-help leaflet on long COVID is distributed, otherwise care as usual by the general practitioner
  Arms: Care as usual and NR; Care as usual and placebo
Dietary Supplement: Placebo — 4 capsules (empty) 2 times daily for 84 days.
  Arms: Care as usual and placebo; MBRT and placebo

SUMMARY:
Long COVID, also referred to as post-acute sequela of COVID-19 (PASC), is present in a substantial number of individuals, and treatment for this is warranted. Two different hypothetical models of Long COVID suggest attenuated mitochondrial energy production and functional brain alterations associated with psychosocial load, respectively, to be key mechanisms in the underlying pathophysiology. Given the potential importance of metabolic disturbances, dietary supplement by Nicotinamide Riboside (NR, sales name Niagen®) may be beneficial. Given the potential importance of functional brain alterations, a tailored and personalized Mind-Body Reprocessing Therapy (MBRT) may be beneficial. The MBRT consists of 4 to 6 face-to-face therapist encounters in combination with digital resources.

The primary objective is to determine whether NR 1000 mg twice daily and/or MBRT increase health-related quality of life in individuals with Long COVID compared with care as usual and/or placebo. The Medical Outcome Study 36-item short form (SF-36), general health subscore is the primary endpoint. Secondary endpoints are: Markers of inflammation (hsCRP) and cognitive function (trail making test), cost-effectiveness, and the patient-reported symptoms fatigue, dyspnoea, and global impression of change in symptoms, function and quality of life. Explorative objectives encompass intervention effects on additional cognitive function markers, biological markers (indices of inflammation and autonomic nervous activity), disability markers (work attendance) and patient symptoms, as well as the exploration of long-term effects, differential subgroup effects, intervention effect mediators and intervention effect predictors.

The study is a randomized controlled trial featuring a 2 x 2 factorial design where MBRT is compared with usual care and NR is compared with placebo. The latter comparison is double blinded. Eligible participants are individuals (18-70 years) with confirmed Long COVID interferring negatively with daily activities. A total of 310 participants will be enrolled. After baseline assessment (T1), the participants will be randomized 1:1 for both treatment comparisons, resulting in four treatment groups: a) MBRT and NR; b) usual care and NR; c) MBRT and placebo; d) usual care and placebo. All treatment periods last for three months, followed by primary endpoint assessment (T2). Total follow-up time is 12 months (T3). A comprehensive investigational program at all time points includes clinical examination, functional testing (spirometry, autonomic cardiovascular control, neurocognitive functions), sampling of biological specimens (blood) and questionnaire charting (background/demographics, clinical symptoms, psychosocial factors, study events).

ELIGIBILITY:
Inclusion Criteria:

* Undergone acute COVID-19, confirmed EITHER by a positive PCR-test OR a positive self-test combined with confirmatory antibody-pattern in blood.
* Persistent symptoms at least 6 months following acute COVID-19 without symptom-free interval.
* Functional disability to an extent that impacts negatively on normal activities (such as work attendance, physical exercise, social activities, etc.)
* Informed consent

Exclusion Criteria:

* Other chronic illnesses, demanding life situations or concomitant drug use/substance abuse that is considered a plausible cause of persistent symptoms and associated disability
* Sustained organ damage (lung, heart, brain) following acute, serious Covid-19
* Pregnancy.
* Bedridden
* Insufficient command of Norwegian

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | Three months after inclusion (T2)
  The Medical Outcome Study 36-item short form (SF-36), general health subscore (total range 0 - 100, where higher scores indicate better QoL)

SECONDARY OUTCOMES:
Inflammation | Three months after inclusion (T2)
  Plasma levels of C-reactive protein, high-sensitive assay (hsCRP). Higher levels indicate more inflammation
Executive functioning | Three months after inclusion (T2)
  The Trail Making test, part B, seconds. Longer time indicates poorer executive functioning
Fatigue | Three months after inclusion (T2)
  Chalder Fatigue Questionnaire (CFQ), total sum score (total range is from 0 - 33; higher scores indicate more fatigue)
Dyspnoea | Three months after inclusion (T2)
  Medical Research Council dyspnoea scale. Total range is from 0 - 4, where higher scores indicate more dyspnoea
Global impression of change | Three months after inclusion (T2)
  Patient Global Impression of Change (PGIC) inventory. Total range is from 1 - 7; higher scores imply that the health status is considered worsened
Cost-effectiveness | Three months after inclusion (T2)
  Incremental cost-effectiveness ratio, using the 36-item short form (SF-36) general health subscore to determine quality-adjusted life years.

OTHER OUTCOMES:
Subjective cognitive difficulties | Three months after inclusion (T2)
  Average score across 4 single items adressing subjective cognitive complaints, each scored on a 1-5 Likert scale. Higher scores means more subjective cognitive difficulties.
Worrying tendencies | Three months after inclusion (T2)
  Penn State Worry Questionnaire (PSWQ), total sum score (higher scores means more worrying)
Sympathetic predominance | Three months after inclusion (T2)
  Heart rate variability (HRV) indices in the time and frequency domain using a 5-minute ECG recording obtained during supine rest
Post-exertional malaise (PEM) | Three months after inclusion (T2)
  PEM items from the DePaul Symptom Questionnaire, total average score across five items
Subjective pain experiences | Three months after inclusion (T2)
  Brief Pain Inventory (BPI), average score
Sleep difficulties | Three months after inclusion (T2)
  Karolinska sleep questionnaire (KSQ), total sum score
Depression | Three months after inclusion (T2)
  Hospital Anxiety and Depression Symptoms (HADS), depression sub-score
Smell and taste abnormalities | Three months after inclusion (T2)
  Averaged score across two singel questionnaire items each scored on a 5-point Likert scale where higher scores means more symptoms
Working memory | Three months after inclusion (T2)
  The digit span test, total score. Higher scores means better working memory
Inflammation, additional information | Three months after inclusion (T2)
  Plasma levels of Interleukin (IL)-6. Higher levels means more inflammation.
Anxiety | Three months after inclusion (T2)
  Hospital Anxiety and Depression Symptoms (HADS), anxiety sub-score
Physical functioning | Three months after inclusion (T2)
  The Medical Outcome Study 36-item short form (SF-36), physical functioning subscore (total range 0 - 100, where higher scores indicate better physical functioning)
Social functioning | Three months after inclusion (T2)
  The Medical Outcome Study 36-item short form (SF-36), social functioning subscore (total range 0 - 100, where higher scores indicate better social functioning)

CONTACTS AND LOCATIONS:
Overall Officials: Torbjørn Omland, PhD, Study Chair — Akershus University Hospital/University of Oslo
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT05703074/Prot_002.pdf
  • Statistical Analysis Plan (2025-02-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT05703074/SAP_004.pdf